CLINICAL TRIAL: NCT06368960
Title: The Study to Evaluate the Safety, PK, and Preliminary Efficacy of BM201 Injection Combined With Radiotherapy in Patients With Unresectable Locally Advanced or Metastatic Solid Tumors That Failed Standard Therapy
Brief Title: BM201 in Combination With Radiotherapy in Patients With Advanced Solid Tumors
Acronym: BM201-1001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: InnoBM Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BM201-1001; CTR20223162 (Registry Identifier: National Medical Products Administration)
Record Dates: First submitted 2024-04-07; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy (Experimental): Radiation：Hypofractionated radiotherapy
  Interventions: Radiation: Radiotherapy
- BM201 injection combined with radiotherapy (Experimental): BM201 injection：Intratumoral injection Radiation：Hypofractionated radiotherapy
  Interventions: Radiation: Radiotherapy; Drug: BM201 injection

INTERVENTIONS:
Radiation: Radiotherapy — Radiation： Hypofractionated radiotherapy
  Other Names: RT
Drug: BM201 injection — BM201 injection：Dose escalation：24mg to 240mg
  Other Names: BM201
  Arms: BM201 injection combined with radiotherapy

SUMMARY:
This is a non-randomized，open-label，controlled multi-center Phase Ⅰ study to evaluate tolerability, pharmacokinetics, and preliminary efficacy of BM201 injection in combination with radiotherapy in patients with histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors who have failed standard therapy or are unable to receive standard treatment.

DETAILED DESCRIPTION:
This is a Phase I, open-label clinical study primarily designed to evaluate the safety and tolerability of BM201 injection in combination with radiotherapy in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable advanced or metastatic solid tumors, either refractory to standard therapy or ineligible for standard treatment.
2. ECOG performance status score of 0-2 point;
3. Expected survival of ≥3 months.
4. At least one measurable lesion by irRECIST criteria, and eligible for intratumoral injection.
5. Prior anti-tumor treatments should be paused for at least 4 weeks before trial initiation，with toxicity related to anti-cancer treatment recovered to ≤Grade 1.
6. Adequate organ and bone marrow function

Exclusion Criteria:

1. Patients with active brain metastasis and/or leptomeningeal carcinomatosis，exempt for asymptomatic brain metastases or stable metastatic lesions for a minimum of 4 weeks.
2. Allergic: History of hypersensitivity to active ingredients or any other components of the study medication; cumulative two or more allergies to contrast agents, other drugs, or food.
3. Active hepatitis B or positive antibodies for hepatitis C, human immunodeficiency virus (HIV), or syphilis.
4. Severe cardiac or cerebrovascular conditions, uncontrolled diabetes, hypertension not well-managed medically (systolic &amp;gt;140 mmHg and/or diastolic &amp;gt;90 mmHg), serious infections (active within 14 days before first drug administration/radiotherapy), active GI ulcers, and immune dysfunction.
5. Presence of other active malignancies or history thereof, except for previously managed non-invasive skin basal or squamous cell carcinomas with a 5-year recurrence-free interval, cervical carcinoma in situ, and ductal carcinoma in situ of the breast.
6. Uncontrolled third-space effusions such as pericardial, abdominal, or pleural within 2 weeks before the initial treatment.
7. Administration of corticosteroids within the preceding 2 weeks before initial treatment.
8. Receipt of vaccination within 2 weeks prior to initial therapy.
9. Participation in clinical trial involving drugs or biologics within 4 weeks before the initial treatment.
10. History of major surgery within 3 months prior to initial treatment or scheduled major surgery during the clinical trial period.
11. Prior blood donation or major hemorrhage (&amp;gt;450 mL) within 3 months before initial therapy, or intention to donate blood/blood components during or within 3 months after the trial.
12. Patients with difficult venous access or intolerance to venipuncture, and those unable to tolerate intratumoral injection.
13. Pregnant (positive pregnancy test) and lactating females.
14. Subjects planning pregnancy or gamete donation within 3 months post-consent and unwilling to practice effective contraception.
15. Patients deemed ineligible for enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT and MTD | Up to 14 days after the initial treatment
  Dose limiting toxicity and maximum tolerated dose
Pharmacokinetic (PK) parameters | From pre-dose to 96 hrs post-dose
  Maximum plasma concentration(Cmax) of the drug after administration
Number of patients with adverse events (AEs) | From the first treatment to 42 days after the last treatment.
  Number of patients with treatment-related adverse events (AEs)

SECONDARY OUTCOMES:
ORR | Up to 42 days after the last treatment
  Objective Response Rate
Peripheral blood cytokine profiling in study participants. | From pre-dose/pre-radiation to 4 hrs post-dose/post-radiation.
  To investigate the change of peripheral blood cytokine level in subjects after the treatment.
The variation in peripheral blood tumor biomarker concentrations. | Up to 42 days after the last treatment
  The variation of concentrations of AFP，NSE，CEA ；
Other exploring outcomes | Up to 14 days after the initial treatment
  The variation of tumor tissue biomarker expression levels

CONTACTS AND LOCATIONS:
Overall Officials: Baorui L Chief Physician, PH.D, Principal Investigator — Nanjing Drum Towel Hospital /The Affiliated Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Towel Hospital /The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No